CLINICAL TRIAL: NCT00824512
Title: Efficacy of EGb761 120mg Bid Versus Placebo in Patients Suffering From Friedreich Ataxia. A 3 Month, Phase II, Randomised, Double Blind, Placebo Controlled, Parallel Group Clinical Study.
Brief Title: Efficacy of EGb761 in Patients Suffering From Friedreich Ataxia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2-39-00240-133; 2007-005371-34 (EudraCT Number)
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2013-05-21 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-03

CONDITIONS: Friedreich Ataxia
MeSH Terms: conditions — Friedreich Ataxia | interventions — Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- EGb 761® 120 mg (Experimental)
  Interventions: Drug: EGb 761 120 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EGb 761 120 mg — EGb 761® 120 mg bid, orally for 12 to 14 weeks
  Arms: EGb 761® 120 mg
Drug: Placebo — Placebo 1 tablet BID, orally for 12 to 14 weeks
  Arms: Placebo

SUMMARY:
The purpose of this protocol is to determine the efficacy of EGb 761 120 mg bid versus placebo in patients suffering from Friedreich Ataxia

ELIGIBILITY:
Inclusion Criteria:

* Friedreich ataxia diagnosis confirmed by evidenced mutation expansion of Frataxin gene
* Ambulatory patient, with depressed tendon reflexes and pyramidal syndrome associated or not to a loss of position or vibration senses or dysarthria
* Patient able to perform the tests of the study

Exclusion Criteria:

* Severe cardiac disease as assessed by echocardiography performed at least within 6 months before screening or during the wash out period (4 weeks)
* Absolute contra-indication to Nuclear Magnetic Resonance spectroscopy(NMR) examination: iron and any magnetic objects implanted in the whole body, e.g. some neurostimulators, cardiac pace-makers, vascular clips and other implanted orthopaedic prosthesis
* Patient who did not deplete at baseline phosphocreatine (PCr) pool by more than 30 % during the exercise bout
* Any continuous use of the following forbidden medications:
* other antioxidant such as idebenone, coenzyme Q, vitamin E/C taken for less than 4 weeks prior study treatment start (ie for antioxidant drugs a mandatory wash-out period of 4 weeks prior study drug start has to be observed),
* any other vasodilators
* tranquilizer such as benzodiazepine, meprobamate or buspirone, and/or antidepressant (only one), at non stable dose

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Hospital Necker Enfants Malades, Paris, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a single centre investigational site in France.
Pre-assignment Details: Overall number of baseline participants differs from number of participants who started as efficacy analysis was performed on modified Intention-To-Treat (mITT) population (i.e. 21 patients). 1 patient in the placebo group did not meet the primary criteria and thus excluded from the analysis. No patient was excluded from the safety population.
Groups:
- EGb 761® 120 mg: EGb 761 120 mg : EGb 761® 120 mg BID, orally for 12 to 14 weeks
- Placebo: Placebo : Placebo 1 tablet BID, orally for 12 to 14 weeks.
Period: Overall Study
Arm/Group | EGb 761® 120 mg | Placebo
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo : Placebo 1 tablet BID, orally for 12 to 14 weeks.
  Baseline Characteristics data is based on the mITT population, which comprised of the 21 patients. One patient in the placebo group was excluded from the analyses because no assessment of the primary criteria was performed.
- Total: Total of all reporting groups
Arm/Group | EGb 761® 120 mg | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Customized [Number; unit: participants]
  12-15 years | 5 | 4 | 9
  16-22 years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 6 | 5 | 11
Duration since first symptoms [Median (Full Range); unit: years] | 8.1 [3 to 15] | 7.7 [4 to 18] | 7.8 [3 to 18]
Number of repeats of Guanine Adenine Adenine (GAA) sequence [Median (Full Range); unit: GAA sequence repetitions] | 700 [500 to 950] | 810 [100 to 1000] | 700 [100 to 1000]

OUTCOME MEASURES:

1. Primary Outcome: Creatine Rephosphorylation Rate Post Exercise
Description: Creatine Rephosphorylation Rate post exercise measured using Phosphorus 31 Nuclear Magnetic Resonance (P-31 NMR)spectroscopy and calculated with correction according to muscular pH.
Time Frame: Baseline (Week 0) to Week 12
Population: Due to small sample size and considering there are no specific studies in this population with EGb761; calculation with the use of a statistical hypothesis was not possible. Primary efficacy analyses performed on the mITT population and analysis of safety performed on the safety population.
Measure: Median (Full Range); unit: pH per second
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
pH per second
  Baseline (Week 0) | 0.024 [0.013 to 0.037] | 0.029 [0.018 to 0.040]
  Week 12 | 0.022 [0.015 to 0.043] | 0.029 [0.014 to 0.035]
  Change from Baseline (Week 0) to Week 12 | 0.001 [-0.009 to 0.009] | 0.000 [-0.013 to 0.005]
Statistical Analysis 1: Comparison: EGb 761® 120 mg vs Placebo; Test type: Superiority or Other; p = 0.9133, Non parametric ANCOVA on the rank test — No multiplicity adjustment performed for this study and all statistical tests are two-sided at the 5% significance level; The baseline value was used as a covariate

2. Secondary Outcome: Peak Post Exercise Perfusion
Description: Peak post exercise perfusion (mL/mn/100 g of tissue) was assessed using Arterial spin labelling combined with Nuclear Magnetic Resonance imaging.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: ml/mn/100 g of tissue
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
ml/mn/100 g of tissue
  Baseline (Week 0) | 54.30 [33.9 to 91.0] | 51.80 [10.8 to 81.4]
  Week 12 | 58.80 [37.6 to 88.8] | 46.60 [30.7 to 63.1]
  Change from Baseline (Week 0) to Week 12 | 3.60 [-29.5 to 31.2] | -1.55 [-20.9 to 23.2]

3. Secondary Outcome: Time to Peak Perfusion
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: seconds
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
seconds
  Baseline (Week 0) | 38.30 [0.8 to 269.3] | 58.55 [5.3 to 317.3]
  Week 12 | 39.80 [0.8 to 119.3] | 76.55 [0.8 to 384.8]
  Change from Baseline (Week 0) to Week 12 | 8.50 [-267.0 to 94.5] | 14.25 [-232.5 to 274.5]

4. Secondary Outcome: Perfusion-time Integral During the First 9 Minutes Post Exercise.
Description: The integral of 'peak perfusion' over a period of 9 minutes post exercise.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: mL/100 g of tissue
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
mL/100 g of tissue
  Baseline (Week 0) | 166.90 [83.6 to 353.0] | 157.20 [11.8 to 373.0]
  Week 12 | 191.60 [86.1 to 417.3] | 185.70 [22.0 to 396.7]
  Change from Baseline (Week 0) to Week 12 | -5.20 [-138.2 to 237.4] | 0.05 [-156.7 to 212.9]

5. Secondary Outcome: Muscle Reoxygenation Rate Post Exercise.
Description: Muscle reoxygenation rate post exercise was assessed using Myoglobin Hydrogen-1 Nuclear Magnetic Resonance spectroscopy.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: per second
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
per second
  Baseline (Week 0) | 0.0870 [0.035 to 0.156] | 0.0540 [0.024 to 0.123]
  Week 12 | 0.0580 [0.030 to 0.114] | 0.0620 [0.021 to 0.087]
  Change from Baseline (Week 0) to Week 12 | -0.0350 [-0.124 to 0.039] | -0.0035 [-0.058 to 0.049]

6. Secondary Outcome: Muscle Trophicity: Maximum Cross Section of Muscle
Description: Muscle trophicity measured using Phosphorus 31 Nuclear Magnetic Resonance (P-31 NMR)spectroscopy and calculated based on maximum cross section of muscle (cm^2)
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: cm^2
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
cm^2
  Baseline (Week 0) | 28.10 [16.6 to 33.1] | 28.95 [23.4 to 42.4]
  Week 12 | 26.8 [16.7 to 33.2] | 29.85 [24.0 to 42.9]
  Change from Baseline (Week 0) to Week 12 | 0.10 [-1.3 to 0.7] | 0.55 [-2.1 to 2.1]

7. Secondary Outcome: Developed Force During the Exercise Bout
Description: Developed force during the exercise bout measured using Phosphorus 31 Nuclear Magnetic Resonance (P-31 NMR)spectroscopy
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Joules
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
Joules
  Baseline (Week 0) | 305.30 [177.0 to 822.9] | 358.10 [207.2 to 1172.8]
  Week 12 | 277.50 [136.90 to 750.9] | 354.35 [200.9 to 1002.1]
  Change from Baseline (Week 0) to Week 12 | -32.40 [-146.9 to 56.6] | 19.20 [-191.8 to 109.8]

8. Secondary Outcome: Normalised Work Developed During the Exercise
Description: Normalised work developed during the exercise was derived as Work developed during the exercise/([60 X Maximum cross section of muscle]-1100).
  Normalised work measured using Phosphorus 31 Nuclear Magnetic Resonance (P-31 NMR)spectroscopy.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: Joules/cm^2
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
Joules/cm^2
  Baseline (Week 0) | 12.07 [6.3 to 26.0] | 12.00 [8.6 to 30.5]
  Week 12 | 9.23 [7.6 to 24.0] | 11.53 [6.1 to 25.7]
  Change from Baseline (Week 0) to Week 12 | -1.03 [-6.3 to 2.6] | 0.47 [-4.8 to 4.6]

9. Secondary Outcome: Metabolism Efficacy Index
Description: The metabolism efficacy index was derived as Normalised work x creatine phosphorylation rate (sec-1). [Normalised work was derived as Work developed during the exercise/(60 X Maximum cross section of muscle-1100)]. Greater values of Metabolism Efficacy index indicate improvement in skeletal muscle energetics while lower values indicate the reverse. Negative values obtained using the formula indicated severe levels of muscle weakness.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: per second
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
per second
  Baseline (Week 0) | 0.0180 [-0.042 to 0.038] | 0.0150 [0.010 to 0.029]
  Week 12 | 0.0130 [-0.021 to 0.042] | 0.0145 [0.007 to 0.028]
  Change from Baseline (Week 0) to Week 12 | 0.0010 [-0.021 to 0.021] | -0.0010 [-0.007 to 0.001]

10. Secondary Outcome: International Cooperative Ataxia Rating Scale [ICARS] (Total Score)
Description: The ICARS was used to measure the general clinical symptoms of Friedreich ataxia using four subscales (i.e. Posture and gait disturbances, Kinetic functions, Speech disorders, & Oculomotor disorders). Scores for each subscale quantify the extent of ataxia in each clinically important area and subscale scores are also summed to give a total score ranging from 0 to 100, with 100 indicative of the most severely affected outcome.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline (Week 0) | 35 [21 to 54] | 26.5 [20 to 58]
  Week 12 | 33.0 [26 to 60] | 29.0 [22 to 54]
  Change from Baseline (Week 0) to Week 12 | 0.0 [-9 to 6] | 0.5 [-4 to 11]

11. Secondary Outcome: ICARS (Posture and Gait Disturbance Score)
Description: The ICARS was used to measure the general clinical symptoms of Friedreich ataxia using four subscales including Posture and gait disturbances. Posture and gait disturbances score range from 0 to 34 (Higher scores indicate higher levels of impairment).
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline (Week 0) | 19.0 [8 to 29] | 12.5 [7 to 31]
  Week 12 | 18.0 [10 to 32] | 12.0 [10 to 29]
  Change from Baseline (Week 0) to Week 12 | 1.0 [-6 to 3] | 2.8 [-3 to 4]

12. Secondary Outcome: ICARS (Kinetic Function Score)
Description: The ICARS was used to measure the general clinical symptoms of Friedreich ataxia using four subscales including Kinetic Function. Kinetic Function score range from 0 to 52 (Higher scores indicate higher levels of impairment).
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline (Week 0) | 15.0 [11 to 19] | 11.5 [9 to 22]
  Week 12 | 13.0 [11 to 24] | 13.0 [11 to 22]
  Change from Baseline (Week 0) to Week 12 | 0.0 [-6 to 5] | 0.5 [-2 to 5]

13. Secondary Outcome: ICARS (Speech Disorders Score)
Description: The ICARS was used to measure the general clinical symptoms of Friedreich ataxia using four subscales including Speech Disorders. Speech Disorders Score range from 0 to 8 (Higher scores indicate higher levels of impairment).
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline (Week 0) | 2.0 [0 to 4] | 0.5 [0 to 3]
  Week 12 | 1.0 [0 to 2] | 1.0 [0 to 2]
  Change from Baseline (Week 0) to Week 12 | 0.0 [-3 to 1] | 0.0 [-1 to 2]

14. Secondary Outcome: ICARS (Oculomotor Disorders Score)
Description: The ICARS was used to measure the general clinical symptoms of Friedreich ataxia using four subscales including Oculomotor Disorders. Oculomotor Disorders score range from 0 to 6 (Higher scores indicate higher levels of impairment).
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
score on a scale
  Baseline (Week 0) | 1.0 [0 to 2] | 1.5 [0 to 3]
  Week 12 | 2.0 [1 to 3] | 2.0 [1 to 2]
  Change from Baseline (Week 0) to Week 12 | 0.0 [0 to 1] | 0.0 [-1 to 2]

15. Secondary Outcome: Timed 25-foot Walk Test
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: seconds
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
seconds
  Baseline (Week 0) | 8.50 [6.0 to 16.0] | 6.75 [5.0 to 29.5]
  Week 12 | 9.00 [7.0 to 15.5] | 6.75 [5.5 to 29.5]
  Change from Baseline (Week 0) to Week 12 | 0.50 [-1.0 to 2.0] | 0.00 [-2.5 to 0.5]

16. Secondary Outcome: Nine Hole Peg Test (Dominant Hand)
Description: The nine hole peg test was used to assess cognitive function and in particular, fine motor coordination. The patient was asked to place nine pegs in nine holes and was scored on the amount of time it took to place and remove all nine pegs.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: seconds
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
seconds
  Baseline (Week 0) | 38.50 [31.5 to 71.5] | 43.50 [33.5 to 91.5]
  Week 12 | 42.00 [29.5 to 86.0] | 40.75 [32.0 to 89.5]
  Change from Baseline (Week 0) to Week 12 | 1.50 [-2.5 to 15.5] | -1.50 [-4.0 to 6.5]

17. Secondary Outcome: Nine Hole Peg Test (Nondominant Hand)
Description: as for outcome 16
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: seconds
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
seconds
  Baseline (Week 0) | 47.50 [39.5 to 113.0] | 48.50 [34.5 to 117.5]
  Week 12 | 53.00 [36.0 to 113.5] | 46.50 [36.5 to 100.5]
  Change from Baseline (Week 0) to Week 12 | 0.50 [-11.0 to 7.0] | 1.75 [-17.0 to 7.0]

18. Secondary Outcome: Choice Reaction Time Test- Reaction Time
Description: The choice reaction time test was used to assess cognitive functioning. On random presentation of one of six signal lights, the patient was asked to respond as quickly and accurately as possible by removing their index finger of the dominant hand from the bottom key and pressing whichever of the top six keys was indicated by the signal. Reaction time was the time elapsed between the presentation of the stimulus and the release of the finger and movement time was defined as the time elapsed between release of the finger and pressure of the second key.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: millisecond
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
millisecond
  Baseline (Week 0) | 513.5 [392 to 1594] | 536.0 [461 to 692]
  Week 12 | 491.0 [417 to 899] | 531.0 [446 to 865]
  Change from Baseline (Week 0) to Week 12 | 8.5 [-1032 to 40] | 9.0 [-89 to 173]

19. Secondary Outcome: Choice Reaction Time Test- Movement Time
Description: as for outcome 18
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: millisecond
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
millisecond
  Baseline (Week 0) | 561.5 [344 to 1452] | 531.0 [390 to 986]
  Week 12 | 555.0 [406 to 1107] | 496.5 [396 to 1419]
  Change from Baseline (Week 0) to Week 12 | 4.5 [-998 to 190] | -31.0 [-124 to 433]

20. Secondary Outcome: Visual Assessment Scale (VAS) of Global Impression - Patient
Description: The VAS used a 10-cm scoring scale in which values were reported in mm such that 0=bad and 100=good. Total score range on VAS is from 0 to 100.
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: mm
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
mm
  Baseline (Week 0) | 60.0 [18 to 80] | 68.5 [12 to 100]
  Week 12 | 67.0 [12 to 82] | 63.0 [26 to 100]
  Change from Baseline (Week 0) to Week 12 | -2.0 [-47 to 30] | -2.0 [-20 to 59]

21. Secondary Outcome: Visual Assessment Scale (VAS) of Global Impression - Parents
Description: as for outcome 20
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: mm
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
mm
  Baseline (Week 0) | 64.0 [45 to 96] | 62.0 [16 to 87]
  Week 12 | 64.0 [31 to 95] | 57.0 [11 to 72]
  Change from Baseline (Week 0) to Week 12 | -7.0 [-14 to 13] | -10.0 [-25 to 14]

22. Secondary Outcome: Visual Assessment Scale (VAS) of Global Impression - Investigator
Description: as for outcome 20
Time Frame: Baseline (Week 0) to Week 12
Population: as for outcome 1
Measure: Median (Full Range); unit: mm
Arm/Group | EGb 761® 120 mg | Placebo
Number analyzed (Participants) | 11 | 10
mm
  Baseline (Week 0) | 78.0 [67 to 90] | 76.0 [25 to 90]
  Week 12 | 80.0 [46 to 87] | 74.0 [46 to 86]
  Change from Baseline (Week 0) to Week 12 | -2.0 [-36 to 13] | -1.0 [-23 to 52]

ADVERSE EVENTS:
Arm/Group | EGb 761® 120 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/11
Other Adverse Events (participants affected / at risk) | 8/11 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGb 761® 120 mg (N=11) | Placebo (N=11)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EGb 761® 120 mg (N=11) | Placebo (N=11)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 1 (1) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Orthopedic procedure (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days